CLINICAL TRIAL: NCT07153419
Title: Cost-Effectiveness and Outcome of Robot-assisted Vs Laparoscopic Roux-en-Y Gastric Bypass: A Non-inferiority Randomized Controlled Trial
Brief Title: Cost-Effectiveness and Outcome of Robot-assisted Vs Laparoscopic Roux-en-Y Gastric Bypass
Acronym: LvRRYGB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5186
Record Dates: First submitted 2023-08-28; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-09

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Laparoscopic RYGB (Active Comparator): Patients undergoing Roux-en-Y gastric bypass (RYGB) surgery performed laparoscopically.
  Interventions: Device: Laparoscopic and robotic (DaVinci) RYGB
- Robotic RYGB (Experimental): Patients undergoing Roux-en-Y gastric bypass (RYGB) surgery performed using the DaVinci robotic platform.
  Interventions: Device: Laparoscopic and robotic (DaVinci) RYGB

INTERVENTIONS:
Device: Laparoscopic and robotic (DaVinci) RYGB — Laparoscopic and robotic (DaVinci) Roux-en-Y Gastric Bypass

SUMMARY:
The objective of this randomized controlled trial is to compare perioperative outcomes between laparoscopic and robotic approaches in patients with severe obesity who are candidates for RYGB. The trial aims to address the following key questions:

To evaluate the difference between the two procedures in terms of postoperative complications.

To assess intraoperative complications, conversion rate, mortality, operative times, postoperative hospital stay, and cost analysis for both approaches.

In summary, the researchers will compare the laparoscopic and robotic approaches to determine which one leads to better perioperative outcomes

DETAILED DESCRIPTION:
Treating patients with pathological obesity has always posed a challenge for bariatric surgeons due to their increased risk of post-operative complications and varying short-term outcomes depending on the chosen procedure. Currently, there are no established guidelines to dictate which procedure is optimal for a given clinical presentation. Surgeons typically make this decision based on their expertise and the patient's characteristics. The most frequently performed procedures worldwide are sleeve gastrectomy and Roux-en-Y gastric bypass, with the latter validated by numerous long-term studies as a safe and effective bariatric and metabolic option for patients with a BMI <50 kg/m2. However, the complexity of Roux-en-Y gastric bypass, which requires the creation of two anastomoses during the reconstruction phase, which might be challenging when performed laparoscopically, may be facilitated by a robotic approach. Although some studies suggest that these approaches have equivalent safety and efficacy profiles, conclusive evidence evaluating their economic impact remains elusive. Consequently, the objective of the present study is to compare morbidity between the laparoscopic and robotic approach in patients undergoing Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients who are candidates for Roux-en-Y gastric bypass using a minimally invasive technique
* Informed consent has been given.

Exclusion Criteria:

* patients who are candidates for bariatric procedures other than Roux-en-Y gastric bypass, or to those who require a laparotomy for Roux-en-Y gastric bypass surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Early complications rate | 30 Days after hospital discharge
  The percentage or proportion of individuals who experience adverse events or negative outcomes within a 30th day of time after hospital discharge

SECONDARY OUTCOMES:
Intraoperative complications rate | From the beginning to the end of the surgical procedure
  The percentage or proportion of individuals who experience adverse events or negative outcomes during surgical procedure.
Conversions rate | From the beginning to the end of the surgical procedure
  The percentage of individuals who start out undergoing a minimally invasive procedure but end up requiring a conversion to a more invasive procedure.
mortality rate | 30 days after hospital discharge
  The percentage or proportion of individuals who die within a 30th day of time after hospital discharge
Operative time | From the beginning to the end of the surgical procedure
  The length of time a patient spends in the operating room undergoing a surgical procedure, from the start of the surgery to the completion of the procedure
Length of hospital stay | up to 1 week
  The amount of time a patient spends in the hospital or medical facility after a surgical procedure has been performed.
Costs of hospitalization and surgery | up to 1 week
  the expenses associated with medical care provided during a patient's stay in a hospital or medical facility, including surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No